CLINICAL TRIAL: NCT03575468
Title: Enhanced E-cigarette Coaching Intervention for Dual Users of Cigarettes and E-cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Collaborators: University of Oklahoma (Other); SRI International (Industry); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DA042960-01A1 (NIH)
Record Dates: First submitted 2018-05-31; First posted 2018-07-02 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Smoking Cessation
Keywords: e-cigarette; vaping; electronic nicotine delivery system (ENDS); smoking cessation
MeSH Terms: conditions — Smoking Cessation; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced E-cigarette Coaching (EEC) (Experimental): The EEC intervention calls will include assessment of e-cigarette use and discussion about how and why e-cigarettes are being used on every call. In addition to the standard quitline cessation program, the enhanced program will include education (via quit coaches and two tailored quit guides), behavioral support tailored to dual users, and shared decision making strategies to address how and why FDA-approved quitting aids and ENDS are being used and to develop an integrated quit plan based on callers' decisions.
  Interventions: Behavioral: Enhanced E-cigarette Coaching
- Quitline treatment as usual (TAU) (Active Comparator): The standard tobacco quitline program is a proactive 5-call intervention grounded in social cognitive theory and the U.S. Public Health Service clinical practices guidelines for treating tobacco use and dependence. All enrollees in the study are eligible for 2-8 weeks of nicotine replacement therapy (depending on their standard quitline benefit offering), if they medically qualify and/or return a medical override letter from their doctor.
  Interventions: Behavioral: Quitline treatment as usual

INTERVENTIONS:
Behavioral: Enhanced E-cigarette Coaching — The EEC intervention calls will include assessment of e-cigarette use and discussion about how and why e-cigarettes are being used on every call. In addition to the standard quitline cessation program, the enhanced program will include education (via quit coaches and two tailored quit guides), behavioral support tailored to dual users, and shared decision making strategies to address how and why FDA-approved quitting aids and ENDS are being used and to develop an integrated quit plan based on callers' decisions.
  Other Names: EEC
  Arms: Enhanced E-cigarette Coaching (EEC)
Behavioral: Quitline treatment as usual — The standard tobacco quitline program is a proactive 5-call intervention grounded in social cognitive theory and the U.S. Public Health Service clinical practices guidelines for treating tobacco use and dependence. All enrollees in the study are eligible for 2-8 weeks of nicotine replacement therapy (depending on their standard quitline benefit offering), if they medically qualify and/or return a medical override letter from their doctor.
  Other Names: TAU
  Arms: Quitline treatment as usual (TAU)

SUMMARY:
The purpose of this study is to develop and pilot test an enhanced behavioral coaching intervention for dual users of cigarettes and electronic nicotine delivery systems (ENDS) who call tobacco quitlines for help quitting smoking.

DETAILED DESCRIPTION:
The specific aims of this research are to:

1. Develop an Enhanced ENDS Coaching (EEC) intervention to improve standard quitline treatment for dual users who contact the quitline for help quitting smoking and are using ENDS, and train tobacco cessation coaches to deliver the intervention.
2. Phase 1 (n=10): Assess preliminary EEC acceptability and feasibility, and refine the intervention with 10 dual users. Hypothesis 1: ENDS users will rate the helpfulness and usability of EEC positively and will exhibit increased knowledge about ENDS and cessation aids.
3. Phase 2 (n=100): Evaluate the feasibility and acceptability of EEC compared to quitline treatment as usual (TAU) in a randomized pilot study of 100 smokers who use ENDS and are seeking help with quitting smoking. Hypothesis 2a (engagement): EEC participants will complete as many or more coaching calls than TAU. Hypothesis 2b (acceptability, satisfaction; assessed via 3-month survey): EEC will have satisfaction at least as high as the TAU group and rate their quit plan development experience more positively. Hypothesis 2c (beliefs; assessed at 3-month survey): EEC participants will report more accurate knowledge and beliefs about ENDS, smoking, and FDA-approved cessation medications.

ELIGIBILITY:
Inclusion Criteria:

* • Requested quitline coaching services and enrolled in 5 call Oklahoma Tobacco Helpline (OKHL) program

  * Currently using e-cigarettes
  * Indicated plan to use e-cigarettes in the next 30 days
  * English Speaking
  * 18+ years old
  * Willing to quit cigarettes in the next 30 days
  * Consented to receive automated phone outreach via the quitline (TCPA consented)
  * Has an Android smartphone with an operating system of 6.0 or higher and comfort downloading and using apps on phone
  * Has regular access to email
  * Callback best time between the hours of 6:00 am - 3:00 pm Pacific Standard Time

Exclusion Criteria:

* • Pregnant or Planning pregnancy within 3 months

  * Reported Schizophrenia diagnosis history during registration
  * Heart attack past 2 weeks
  * Stroke/Transient Ischemic Attack past 2 weeks
  * Rapid Irregular heart beat past 6 months
  * Angina or heart pain past 6 months
  * Currently taking Varenicline (also known as Chantix) or Bupropion (also known as Wellbutrin or Zyban)
  * Previously screened for study
  * Enrolled via proxy (i.e., did not self-enroll)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Vickerman, PHD, Principal Investigator — Optum, Inc.
Locations (1):
- Optum, Seattle, Washington, United States

REFERENCES:
- [Result] Vickerman KA, Carpenter KM, Miles LN, Hsu JM, Watt KA, Brandon TH, Hart JT, Javitz HS, Wagener TL. Treatment development, implementation, and participant baseline characteristics: A randomized pilot study of a tailored quitline intervention for individuals who smoke and vape. Contemp Clin Trials Commun. 2021 Sep 8;24:100845. doi: 10.1016/j.conctc.2021.100845. eCollection 2021 Dec. PMID 34568637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Started | 56 | 54
Completed | 30 | 33
Not Completed | 26 | 21
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Call 1 completion required to stay in study per consent process (not contacted for 3-month survey) | 10 | 4
Not completed — Lost to Follow-up | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 46 | 50 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 47 | 90
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 16 | 21 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 12
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 32 | 30 | 62
  More than one race | 4 | 11 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 50 | 96

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction and Acceptability Measured on a Scale From 1-6 (Very Satisfied to Very Dissatisfied)
Description: In Phase 2, average treatment satisfaction and acceptability rating will be compared for EEC and TAU participants. Full 1-6 scale description: 1 - very satisfied; 2 - satisfied; 3 - somewhat satisfied; 4 - somewhat dissatisfied; 5 - dissatisfied; 6 - very dissatisfied. Participants can also respond "I don't know" or "I prefer not to answer". On scale 1-6, 1 is the best outcome.
Time Frame: 3 months after baseline
Population: This analysis focused on 3-month survey respondents (N=66).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Number analyzed (Participants) | 32 | 34
units on a scale | 5.5 [5.3 to 5.8] | 5.0 [4.5 to 5.5]

2. Primary Outcome: Treatment Engagement: Call Completion
Description: In Phase 2, call completion (captured via standard quitline data systems) will be compared for EEC and TAU participants. There is no limit to number of calls that can be completed, although participants are called to complete 5 scheduled calls (best outcome).
Time Frame: Phase 2 time frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: Coaching calls completed
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Number analyzed (Participants) | 32 | 34
Coaching calls completed | 3.4 (.24) | 2.7 (.19)

3. Secondary Outcome: Quit Plan Development Experience
Description: In Phase 2, quit plan development experience will be compared for EEC and TAU participants. Quit plan development experience will be measured with an adapted version of the CollaboRATE (not an abbreviation) shared decision making assessment measure. The adapted CollaboRATE measure included 3 questions (on a 5-point scale from "no effort (0)" to "every effort was made (4)"): "How much effort was made to help you understand your options for quitting smoking?", "How much effort was made to listen to the things that matter most to you about your plan for quitting smoking?", and "How much effort was made to include what matters most to you in creating your plan for quitting smoking?". Higher total scores indicate greater utilization of a shared decision-making approach during quit plan development. Scale minimum equals 0 and maximum equals 12.
Time Frame: 3 months after baseline
Population: Analysis focused on 3-month survey respondents (N=66).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Number analyzed (Participants) | 32 | 34
score on a scale | 10.0 (0.4) | 9.2 (0.6)

4. Secondary Outcome: Knowledge and Beliefs- Relative Risk of ENDS and Cigarettes
Description: In Phase 2, Knowledge and Beliefs about ENDS, Smoking, and FDA-approved Cessation Medications was assessed via 3 relative risk questions about ENDS, Smoking, and FDA-approved Cessation Medications designed for this study, and compared for EEC and TAU participants. Responses to individual items will be described. To assess the relative risk of ENDS and cigarettes, the following question was asked, "Compared to cigarettes, how harmful are e-cigarettes to a person's health?" Answer responses included: less harmful, about the same, more harmful, and I prefer not to answer.
Time Frame: Phase 2 time frame: 3 months after baseline
Population: Respondents to the 3-month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Number analyzed (Participants) | 30 | 33
Participants
  Less Harmful | 22 | 22
  About the Same | 6 | 5
  More Harmful | 0 | 5
  I prefer not to answer | 2 | 1

5. Other Pre Specified Outcome: 7-Day Point Prevalence Smoking Cessation Rates
Description: In Phase 2 participants will report their quit status during their outcome survey.
Time Frame: Phase 2 time frame: 3 months after baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Use of ENDS, Nicotine Replacement Therapy (NRT), and Cigarettes
Description: A descriptive analysis of how ENDS, NRT, and cigarettes are used during a participant's quit process through diary procedures.
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Knowledge and Beliefs- Relative Risk of FDA-approved Cessation Medications and Cigarettes
Description: In Phase 2, Knowledge and Beliefs about ENDS, Smoking, and FDA-approved Cessation Medications was assessed via 3 relative risk questions about ENDS, Smoking, and FDA-approved Cessation Medications designed for this study, and compared for EEC and TAU participants. Responses to individual items will be described. To assess the relative risk of FDA-approved Cessation Medications and cigarettes, the following question was asked, "Compared to cigarettes, how harmful are quit medications like the nicotine patch to a person's health?" Answer responses included: less harmful, about the same, more harmful, and I prefer not to answer.
Time Frame: Phase 2 time frame: 3 months after baseline
Population: Respondents to the 3-month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Number analyzed (Participants) | 30 | 33
Participants
  Less Harmful | 25 | 32
  About the Same | 1 | 1
  More Harmful | 1 | 0
  I Prefer Not to Answer | 3 | 0

8. Secondary Outcome: Knowledge and Beliefs- Relative Risk of FDA-approved Cessation Medications and ENDS
Description: In Phase 2, Knowledge and Beliefs about ENDS, Smoking, and FDA-approved Cessation Medications was assessed via 3 relative risk questions about ENDS, Smoking, and FDA-approved Cessation Medications designed for this study, and compared for EEC and TAU participants. Responses to individual items will be described. To assess the relative risk of FDA-approved Cessation Medications and ENDS, the following question was asked, "Compared to quit medications like the nicotine patch, how harmful are e-cigarettes to a person's health?" Answer responses included: less harmful, about the same, more harmful, and I prefer not to answer.
Time Frame: Phase 2 time frame: 3 months after baseline
Population: Respondents to the 3-month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
Number analyzed (Participants) | 30 | 33
Participants
  Less Harmful | 12 | 4
  About the Same | 5 | 9
  More Harmful | 10 | 19
  I Prefer Not to Answer | 3 | 1

ADVERSE EVENTS:
Time Frame: Outcomes surveys were completed approximately 3-months after baseline and randomization.
Description: Only participants who responded to the 3-month survey and reported use of e-cigs and/or NRT were assessed for Other (Not Including Serious) Adverse Events. Participants who reported use of e-cigs or NRT since study enrollment were asked whether they experienced any side effects related to (1) using e-cigs (if they reported use) and (2) related to using NRT (if they reported use) using two separate questions. Participants could be at risk for adverse events related to both NRT and e-cig use.
Arm/Group | Enhanced E-cigarette Coaching (EEC) | Quitline Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/50
Other Adverse Events (participants affected / at risk) | 17/30 | 19/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Enhanced E-cigarette Coaching (EEC) (N=30) | Quitline Treatment as Usual (TAU) (N=33)
Sore throat d/t reported use of e-cigarette (Respiratory, thoracic and mediastinal disorders) | 9/26 | 4/26
Headache d/t reported use of e-cigarettes (General disorders) | 6/26 | 1/26
Breathing difficulties d/t reported e-cigarette use (General disorders) | 3/26 | 4/26
Cough d/t reported e-cigarette use (Respiratory, thoracic and mediastinal disorders) | 3/26 | 2/26
Dizziness d/t reported e-cigarette use (General disorders) | 3/26 | 2/26
Bad or vivid dreams/nightmares d/t reported e-cigarette use (General disorders) | 3/26 | 1/26
Nausea/stomach upset d/t reported e-cigarette use (General disorders) | 2/26 | 1/26
Chest pain d/t reported e-cigarette use (General disorders) | 1/26 | 2/26
Skin Irritation - rash, itchiness d/t reported NRT use (General disorders) | 2/25 | 2/30
Headache d/t reported NRT use (General disorders) | 3/25 | 2/30
Nausea/stomach upset d/t reported NRT use (General disorders) | 1/25 | 6/30
Any side effect d/t reported e-cigarette use (General disorders) | 14/26 | 11/26
Any side effect d/t NRT use (General disorders) | 10/25 | 12/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT03575468/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03575468/SAP_001.pdf